CLINICAL TRIAL: NCT03380845
Title: Comparison of Fractional Erbium-Doped 1,550-nm Laser and a Bipolar Fractional Radiofrequency Microneedle Device for the Treatment of Atrophic Acne Scars in Ethnic Skin: A Randomized Split-Face Controlled Pilot Study
Brief Title: Comparison of 1,550-nm Laser and Fractional Radiofrequency Microneedle for the Treatment of Acne Scars in Ethnic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Society for Dermatologic Surgery (Other)
Responsible Party: Principal Investigator, Mathew Avram, MD, JD, Director, MGH Laser, Cosmetic and Dermatologic Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P002061
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acne Scars

STUDY DESIGN:
Intervention Model Description: Randomized split-face clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fraxel Restore on one side of the face (Active Comparator): Fraxel Restore on one side of the face
  Fraxel Restore: acne scar correction
  Randomized treatment with Fraxel Restore on one side of the face, and Fractora on the opposite side of the face - the study is a randomized,single-center, split-face study in subjects seeking acne scar correction. Subjects were treated with Fraxel on one side of the face and Fractora on the other side of the face. The side of the face for each device was randomly assigned.
  Interventions: Device: Fraxel Restore
- Fractora on the other side of the face (Active Comparator): Fractora on the other side of the face
  Fractora: acne scar correction
  Randomized treatment with Fraxel Restore on one side of the face, and Fractora on the opposite side of the face - the study is a randomized,single-center, split-face study in subjects seeking acne scar correction. Subjects were treated with Fraxel on one side of the face and Fractora on the other side of the face. The side of the face for each device was randomly assigned.
  Interventions: Device: Fractora

INTERVENTIONS:
Device: Fraxel Restore — Non-ablative Laser. In the study, one side of the face will be treated with Fraxel Restore monthly for three months.
  Arms: Fraxel Restore on one side of the face
Device: Fractora — Fractional Radiofrequency Microneedling Device. In the study, one side of the face will be treated with Fractora monthly for three months.
  Arms: Fractora on the other side of the face

SUMMARY:
The primary objective of this randomized, split-face, controlled study is to compare the efficacy and safety of a erbium-doped 1,550-nm non-ablative fractional laser and a bipolar fractional radiofrequency microneedle device for the treatment of atrophic facial acne scars in ethnic skin (Fitzpatrick Skin Phototypes III-VI).

The hypothesis of this study is that both erbium-doped 1,550-nm non-ablative fractional laser and the bipolar fractional radiofrequency microneedle device are equally effective for the treatment of atrophic acne scars in ethnic skin (SPT III-VI). However, the bipolar fractional radiofrequency microneedle device has less adverse effects than erbium-doped 1,550-nm non-ablative fractional laser due to the absence of scattering and the absence of chromophore-specific targets - predominantly melanin - traditionally needed with laser treatments; hence the fractional radiofrequency microneedle device will have a higher safety profile in darker skin types .

DETAILED DESCRIPTION:
Acne is a highly prevalent disease and post-acne scaring has shown to have detrimental effects on a person's physical, mental, and social well-being. Acne scars can be divided in general categories of hypertrophic or keloid scars, atrophic scars (icepick, rolling, boxcar), and pigmentation alterations (redness, hypo and hyper-pigmentation). This study will focus on treatment of moderate to severe grades of atrophic acne scarring. Our aim is to compare the efficacy and safety of a erbium-doped 1,550-nm non-ablative fractional laser and a bipolar fractional radiofrequency microneedle device for the treatment of atrophic acne scars in ethnic skin (Fitzpatrick Skin Phototypes III-VI) by performing a split-face randomized controlled trial.

Both devices in this study are already FDA approved treatment modalities for acne scarring.

History of erbium-doped 1,550-nm non-ablative fractional laser (Fraxel® Restore Laser System, Solta Medical, Inc., Hayward, CA):

Non-ablative fractional lasers work via the theory of fractional photothermolysis, which creates hundreds to thousands of microscopic thermal zones (MTZs), or columns of thermally injured skin, while sparing the surrounding tissue. The pixilated nature of treatment and the functionally unimpaired stratum corneum allow for rapid tissue healing and allows for safer treatments of our patients. Mechanistically, fractional photothermolysis allows controlled amounts of high energy to be delivered deep within the dermis resulting in collagenolysis and neocollagenesis, which smoothes the textural abnormalities of acne scarring.

Multiple published studies have demonstrated that erbium-doped 1,550-nm non-ablative fractional laser ("NAFL") can be successfully utilized in the treatment of all forms of atrophic acne scarring - ice-pick, boxcar, and rolling scars - with a very favorable safety profile in all skin types, and thus, has been cleared by Food and Drug Administration (FDA) for that particular indication. According to the manufacture manual (reference attached in the "Attachments" section), NAFL is indicated for "use in skin resurfacing procedures as well as treatment of acne scars, surgical scars, lentigos (age spots), solar lentigos (sun spots), actinic keratosis, and melasma."

History of the fractional radiofrequency microneedle device (Fractora; Invasix Ltd./InMode MD Ltd., Israel):

Fractional radiofrequency is not a laser. Instead, these devices use an array of electrodes that allows for zones of thermal wounds to be created between areas of unaffected zones, thus stimulating dermal remodeling and allowing for a supply of reservoir cells to promote healing. Variations of fractional radiofrequency exist that employ microneedles to deliver electrical current to a particular depth within the dermis that decreases damage to the epidermis. These fractional radiofrequency microneedle devices provide an alternative to conventional methods of acne-scar treatment (such as NAFL). Great interest has been culminating over the recent years for the use of such devices in acne scars due to the absence of light scattering and the absence of chromophore-specific targets traditionally needed with laser treatments. As melanin is not a target, it is felt to have a higher safety profile in darker skin phototypes.

A recent study investigated the safety and efficacy of a specific bipolar fractional radiofrequency microneedle device (Fractora; Invasix Ltd./InMode MD Ltd., Israel) for acne and acne scarring. In this study, 8 patients with acne scars were reported and it was noted that all patients (regardless of their skin phototypes) had improvement in their active acne and acne scars after 4 treatments and a 1 month, on average follow-up period. The treatment was well tolerated without any side-effects. Skin biopsies from this study showed reduction in scar depth and new collagen formation with an increase in elastic fibers and adnexal structures noted. A follow-up report showed that 4 out of 8 patients who were in the original study returned for a long term follow-up from 1 to 2 years, that showed ongoing clinical improvements in these patients. This specific bipolar fractional radiofrequency microneedle ("FRM") device has been FDA-approved for acne scars and skin rejuvenation.

To this date the efficacy and safety of 1,550-nm fractionated photothermolysis system has not been compared to a fractional radiofrequency microneedle device for atrophic acne scars in ethnic skin in a randomized split-face controlled trial. A major advantage of a split-face self-controlled design would be to minimize any confounding factors. Laser resurfacing has been well studied and is widely used in individuals with fair skin - Fitzpatrick skin phototypes (SPT) I to II. However, there is a paucity of published studies involving individuals with darker skin types (SPT III-VI)-a population that has a higher risk of laser-associated dyspigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with Fitzpatrick skin types III through VI and facial acne scarring of grades III-IV will be enrolled. Both sides of the participants' face should have almost similar amount and severity of acne scarring. Participants will be over 18 years old

Exclusion Criteria:

* Patients have to be overall healthy without a history of keloidal scarring, localized or active infection in the treatment region, immunodeficiency disorders, porphyria or light sensitivity, and connective tissue disorders. Per PI discretion, any serious medical condition that may interfere with the study. In addition, pregnant or nursing women, patients who have been taking isotretinoin for a period of 6 months before treatment, and patients who have received any cosmetic treatment (lasers, dermabrasion, chemical peels, etc) in the previous 6 months will be excluded. Also, patients with renal disease, and any allergies to Lidocaine, Tetracaine, or Valtrex will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Avram, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Purvis D, Robinson E, Merry S, Watson P. Acne, anxiety, depression and suicide in teenagers: a cross-sectional survey of New Zealand secondary school students. J Paediatr Child Health. 2006 Dec;42(12):793-6. doi: 10.1111/j.1440-1754.2006.00979.x. PMID 17096715
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Alster TS, Tanzi EL, Lazarus M. The use of fractional laser photothermolysis for the treatment of atrophic scars. Dermatol Surg. 2007 Mar;33(3):295-9. doi: 10.1111/j.1524-4725.2007.33059.x. PMID 17338686
- [Background] Chrastil B, Glaich AS, Goldberg LH, Friedman PM. Second-generation 1,550-nm fractional photothermolysis for the treatment of acne scars. Dermatol Surg. 2008 Oct;34(10):1327-32. doi: 10.1111/j.1524-4725.2008.34284.x. PMID 19040687
- [Background] Mahmoud BH, Srivastava D, Janiga JJ, Yang JJ, Lim HW, Ozog DM. Safety and efficacy of erbium-doped yttrium aluminum garnet fractionated laser for treatment of acne scars in type IV to VI skin. Dermatol Surg. 2010 May;36(5):602-9. doi: 10.1111/j.1524-4725.2010.01513.x. Epub 2010 Apr 1. PMID 20384757
- [Background] Alexis AF, Coley MK, Nijhawan RI, Luke JD, Shah SK, Argobi YA, Nodzenski M, Veledar E, Alam M. Nonablative Fractional Laser Resurfacing for Acne Scarring in Patients With Fitzpatrick Skin Phototypes IV-VI. Dermatol Surg. 2016 Mar;42(3):392-402. doi: 10.1097/DSS.0000000000000640. PMID 26945321
- [Background] Hruza G, Taub AF, Collier SL, Mulholland SR. Skin rejuvenation and wrinkle reduction using a fractional radiofrequency system. J Drugs Dermatol. 2009 Mar;8(3):259-65. PMID 19271373
- [Background] Chandrashekar BS, Sriram R, Mysore R, Bhaskar S, Shetty A. Evaluation of microneedling fractional radiofrequency device for treatment of acne scars. J Cutan Aesthet Surg. 2014 Apr;7(2):93-7. doi: 10.4103/0974-2077.138328. PMID 25136209
- [Background] Chae WS, Seong JY, Jung HN, Kong SH, Kim MH, Suh HS, Choi YS. Comparative study on efficacy and safety of 1550 nm Er:Glass fractional laser and fractional radiofrequency microneedle device for facial atrophic acne scar. J Cosmet Dermatol. 2015 Jun;14(2):100-6. doi: 10.1111/jocd.12139. Epub 2015 Mar 23. PMID 25810322
- [Background] Abdel Hay R, Shalaby K, Zaher H, Hafez V, Chi CC, Dimitri S, Nabhan AF, Layton AM. Interventions for acne scars. Cochrane Database Syst Rev. 2016 Apr 3;4(4):CD011946. doi: 10.1002/14651858.CD011946.pub2. PMID 27038134

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: side of the face treated
Groups:
- Bilateral Facial Treatment With Fraxel and Fractora: Randomized treatment with Fraxel on one side of the face, and Fractora on the opposite side of the face - the study is a randomized, split-face study in subjects seeking facial acne scar correction. Subjects were treated with Fraxel on one side of the face and Fractora on the other side of the face. The side of the face for each device was randomly assigned.
Period: Overall Study
Arm/Group | Bilateral Facial Treatment With Fraxel and Fractora
Started | 4; 8 side of the face treated (Participants got bilateral face treatments with Fraxel on one side of face; Fractora on the other.)
Completed | 4; 8 side of the face treated
Not Completed | 0; 0 side of the face treated

BASELINE CHARACTERISTICS:
Population: There were 4 participants enrolled and treated, the participants received bilateral facial treatments with Fraxel on one side of the face, and Fractora on the other side of the face.
Units Other Than Participants: side of the face treated
Groups:
- Split Face Study Bilateral Fraxel Restore vs Fractora: Randomized treatment with Fraxel Restore on one side of the face, and Fractora on the opposite side of the face - the study is a randomized,single-center, split-face study in subjects seeking acne scar correction. Subjects were treated with Fraxel on one side of the face and Fractora on the other side of the face. The side of the face for each device was randomly assigned.
Arm/Group | Split Face Study Bilateral Fraxel Restore vs Fractora
Number analyzed (Participants) | 4
Number analyzed (side of the face treated) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Fitzpatrick Skin Type (FST) Classification [Count of Participants; unit: Participants] — FST Type I skin always burns, never tans (pale white; blond or red hair; blue, gray eyes; freckles) FST Type II skin usually burns, tans minimally (white; blond, brown or red hair; blue, green, or hazel eyes) FST Type III skin sometimes has a mild burn, tans uniformly (cream white; yellowish; any hair color or brown eyes) FST Type IV skin burns minimally, always tans well (light brown; olive; dark brown to black hair) FST Type V skin very rarely burns, tans very easily (brown) FST Type VI skin never burns, always tans (deeply pigmented dark brown to darkest brown, black in complexion)
  Participants
    FST III | 3
    FST VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Acne Scarring - From Baseline to Three Months After Last Treatment
Description: Improvement in acne scarring will be measured by two blinded evaluators both by in-person assessments and by photographic review (digital photography will be used under standardized conditions). A quartile grading scale (1 = 1% to 25%, 2 =26% to 50%, 3 =51% to 75%, 4 = >76% improvement) will be used to measure acne scar improvement. Higher score means better outcome.
Time Frame: three months after last treatment
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: side of face treated
Groups:
- Fraxel Restore on One Side of the Face: Fraxel Restore on one side of the face for acne scar correction
- Fractora on Other Side of the Face: Fractora on other side of the face for acne scar correction
Arm/Group | Fraxel Restore on One Side of the Face | Fractora on Other Side of the Face
Number analyzed (Participants) | 4 | 4
Number analyzed (side of face treated) | 4 | 4
score on a scale | 2 [1 to 3] | 2 [1 to 3]

2. Secondary Outcome: Comparing Side Effects of the Different Lasers
Description: measure side effects by patient reported adverse events and blinded physician assessment of adverse effects. Parameters, include erythema, edema, blistering, crusting, scarring, hypopigmentation, and hyperpigmentation, will be graded on a 4-point scale (0 = absent, 1= mild, 2 = moderate, and 3 = severe). Higher score means worse outcome.
Time Frame: treatment visit 1, treatment visit 2, treatment visit 3, three months after last treatment
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: side of face treated
Arm/Group | Fraxel Restore on One Side of the Face | Fractora on Other Side of the Face
Number analyzed (Participants) | 4 | 4
Number analyzed (side of face treated) | 4 | 4
score on a scale | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Comparing Intensity of Pain With the Different Lasers
Description: Patients will also be evaluated the intensity of pain using a visual analogue scale (0 = absence of pain, 10 = most-severe pain). Higher score means worse outcome
Time Frame: treatment visit 1, treatment visit 2, treatment visit 3
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: side of face treated
Arm/Group | Fraxel Restore on One Side of the Face | Fractora on Other Side of the Face
Number analyzed (Participants) | 4 | 4
Number analyzed (side of face treated) | 4 | 4
score on a scale | 3 [2 to 5] | 7 [6 to 8]

ADVERSE EVENTS:
Time Frame: 6 months
Description: measure adverse events by patient reported adverse events and blinded physician assessment of adverse effects on follow up visits 4 weeks after each treatment as well as at final follow up 3 months after last treatment.
Arm/Group | Fraxel Restore on One Side of the Face | Fractora on Other Side of the Face
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03380845/Prot_SAP_000.pdf